CLINICAL TRIAL: NCT04009161
Title: Osteoradionecrosis Rate in Patients Undergoing Radiotherapy for Head and Neck Cancer Treatment: a Perspective Clinical Study.
Brief Title: Osteoradionecrosis Rate in Patients Undergoing Radiotherapy for Head and Neck Cancer Treatment.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Principal Investigator, Catholic University of the Sacred Heart
Other Study IDs: ORN-HN-1
Record Dates: First submitted 2019-06-19; First posted 2019-07-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer; Osteoradionecrosis; Radiotherapy Side Effect; Tooth Avulsion
MeSH Terms: conditions — Head and Neck Neoplasms; Osteoradionecrosis; Radiation Injuries; Tooth Avulsion | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tooth extraction — Tooth extraction before the beginning of radiotherapy in patients irradiated for Head and Neck cancer

SUMMARY:
Objectives High-dose radiotherapy (RT) for head and neck cancer has significant adverse effects on maxillofacial tissues, among which osteoradionecrosis (ORN) is the most severe and potentially life-threatening. Although tooth extractions seem to be the main risk factor, few perspective studies evaluated protocols to minimize the ORN risk due to extractions. The aim of this study is to evaluate incidence and risk factors of ORN in a cohort of patients receiving tooth extractions before RT and evaluate an algorithm about extraction decision.

Methods One-hundred ten patients were consecutively recruited in this study: impacted third molars with radiographic sign of pericoronitis, teeth with periapical lesions, unrestorable teeth, periodontally compromised teeth (pocket probing depth >5 mm, clinical attachment loss > 8 mm, grade 2 tooth mobility, II grade furcation involvement) were extracted under antibiotic prophylaxis. A 15-days interval between the last tooth extraction and the beginning of RT was recommended. Patients were visited at 15 days, 1, 3 and 6 months after the beginning of RT. Data of patients with a minimum of 6 months follow-up are presented in this report. ORN was defined as irradiated exposed necrotic bone, without healing for 3 months, in absence of cancer recurrence. The protocol was approved by the Ethic Committee of Catholic University - Fondazione Policlinico Gemelli (Prot. OHHN-1, ID-2132).

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the informed consent form
* Patients with diagnosis of HNC, with specific prescription of local radiotherapy, both for curative and palliative purpose, with or without chemotherapic treatment.
* Patient with diagnosis of HNC, with specific prescription of local radiotherapy as an adjuvant to surgical resection, with or without chemotherapic treatment.

Exclusion Criteria:

* Patients participating to other clinical studies
* Patients who refuse to participate in the study
* Patients unable to attend the ambulatory visits scheduled by the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients irradiated for head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Osteoradionecrosis Incidence | 60 months after the beginning of RT
  To evaluate the ORN incidence in a population irradiated for Head and Neck Cancer.
Osteoradionecrosis rate following pre-radiotherapy tooth extraction | 60 months after the beginning of RT

SECONDARY OUTCOMES:
Extraction site: number of tooth extractions for each site (anterior and posterior maxilla or mandible and specific tooth number) and percentage of ORN for each site. | 60 months after the beginning of RT
  Risk of ORN per extraction site
Time interval between extraction and Radiotherapy: days between every tooth extraction and the beginning of RT. | 60 months after the beginning of RT
  To understand the relationship between this time-lapse and the ORN incidence
Surgical protocol 1: Flap elevation per each extracted tooth (YES/NO) and percentage of ORN per each type of procedure. | 60 months after the beginning of RT
  Tooth extraction related risk factors
Surgical protocol 2: Primary intention closure achievement per post-extractive site (YES/NO) and percentage of ORN per each type of procedure. | 60 months after the beginning of RT
  Tooth extraction related risk factors
Surgical protocol 3: Osteotomy per each extracted tooth (YES/NO) and percentage of ORN per each type of procedure. | 60 months after the beginning of RT
  Tooth extraction related risk factors
Reason for tooth extraction: number of tooth extraction for each cause under the protocol (caries, periodontal disease, endodontic lesions, pericoronitis, fracture) and percentage of ORN for each cause. | 60 months after the beginning of RT
  Tooth extraction related risk factors
Radiation dose to the post-extractive site (Gy of radiation received by every post-extractive site) | 60 months after the beginning of RT
  Tooth extraction related risk factors
Age of every patients at the beginning of RT | At baseline
  ORN risk factors
Sex (male, female) of every patients at the beginning of RT | At baseline
  ORN risk factors
Number of participants undergoing concurrent chemotherapy (neoadjuvant or concomitant) | During treatment
  ORN risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rupe C, Gioco G, Massaccesi M, Tagliaferri L, Pastore F, Micciche F, Galli J, Mele D, Specchia ML, Cassano A, Cordaro M, Lajolo C. Osteoradionecrosis incidence in pre-radiation teeth extractions: A prospective study. Oral Dis. 2024 Nov;30(8):5129-5139. doi: 10.1111/odi.14941. Epub 2024 Apr 9. PMID 38591808
- [Derived] Rupe C, Gioco G, Almadori G, Galli J, Micciche F, Olivieri M, Cordaro M, Lajolo C. Oral Candida spp. Colonisation Is a Risk Factor for Severe Oral Mucositis in Patients Undergoing Radiotherapy for Head & Neck Cancer: Results from a Multidisciplinary Mono-Institutional Prospective Observational Study. Cancers (Basel). 2022 Sep 29;14(19):4746. doi: 10.3390/cancers14194746. PMID 36230669